CLINICAL TRIAL: NCT02748395
Title: Lidocaine and Triamcinolone vs Saline Trigger Point Injection for Treatment of Chronic Abdominal Wall Pain
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No IRB approval
Sponsor: Temple University (Other)
Responsible Party: Principal Investigator, Adam Ehrlich, Assistant Professor of Medicine, Temple University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 23417
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Abdominal Wall Pain; Abdominal Cutaneous Nerve Entrapment Syndrome
MeSH Terms: interventions — Triamcinolone; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Injection of 3.5mL of normal saline into the point of maximal tenderness in the abdomen
  Interventions: Other: Placebo
- Treatment (Experimental): Injection of 20mg triamcinolone and 1% lidocaine into the point of maximal tenderness in the abdomen
  Interventions: Drug: Triamcinolone; Drug: Lidocaine

INTERVENTIONS:
Drug: Triamcinolone
  Arms: Treatment
Other: Placebo
  Arms: Placebo
Drug: Lidocaine
  Arms: Treatment

SUMMARY:
The purpose of this study is to determine whether the injection of triamcinolone and lidocaine is effective in relieving chronic abdominal wall pain.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic abdominal wall pain
* Prior ultrasound or cross-sectional imaging of the abdomen to exclude other causes
* Baseline Brief Pain Inventory score ≥ 5

Exclusion Criteria:

* Multiple trigger points
* Abdominal wall hernia on exam
* Weight loss
* Rectal bleeding
* Recent change in bowel habits
* Decompensated cirrhosis or recurrent ascites
* Allergy or contraindication to study medications
* Known thrombocytopenia with platelet count < 50,000
* Other diagnosis of chronic pain syndromes including fibromyalgia
* Unable to provide informed consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pain score | Baseline and 1 month
  Questionnaire to assess change in pain score

SECONDARY OUTCOMES:
Pain score | Baseline and 1 week
  Questionnaire to assess change in pain score
Pain score | Baseline and 2 months
  Questionnaire to assess change in pain score

IPD SHARING:
Plan to Share IPD: Undecided